CLINICAL TRIAL: NCT07073833
Title: An Open Label, Multicenter Phase I Clinical Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of IBR900 Cell Injection in the Treatment of Relapsed/Refractory CD20 Positive B-cell Non Hodgkin Lymphoma
Brief Title: The Safety, Tolerability, and Efficacy of IBR900 Cell Injection in Relapsed/Refractory B-cell Non Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Imbioray (Hangzhou) Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IBR900-101
Record Dates: First submitted 2025-06-26; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ia，single-agent dose escalation of IBR900 cell injection (Experimental)
  Interventions: Drug: IBR900 cell injection
- Phase Ib，monotherapy expansion (queue 1) (Experimental)
  Interventions: Drug: IBR900 cell injection
- Phase Ib，combination expansion (queue 2) (Experimental)
  Interventions: Drug: IBR900 cell injection; Drug: rituximab

INTERVENTIONS:
Drug: IBR900 cell injection — NK cells
Drug: rituximab — CD20 antibody
  Arms: Phase Ib，combination expansion (queue 2)

SUMMARY:
This is an open label clinical study: Phase Ia is a dose escalation phase, evaluating the safety, tolerability, RP2D, PK characteristics, and preliminary efficacy of IBR900 cell injection in the treatment of relapsed/refractory B-cell non Hodgkin lymphoma (NHL); Phase Ib is the dose expansion stage, which is divided into two parts: monotherapy expansion (queue 1) and combination expansion (queue 2). The monotherapy expansion part evaluates the safety, tolerability, and preliminary efficacy of IBR900 cell injection in the treatment of relapsed/refractory CD20 positive B-cell non Hodgkin lymphoma, while the combination expansion part evaluates the safety, tolerability, and preliminary efficacy of IBR900 cell injection combined with CD20 monoclonal antibodies in the treatment of relapsed/refractory CD20 positive B-cell non Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form, understand the study and be willing to follow the protocol and complete all experimental procedures;
2. Male or female, age ≥ 18 years old;
3. CD20 positive B-cell non Hodgkin's lymphoma (B-NHL), including but not limited to diffuse large B-cell lymphoma non-specific, high-grade B-cell lymphoma with MYC and BCL2 rearrangements, high-grade B-cell lymphoma with MYC/BCL2/BCL6 rearrangements, high-grade B-cell lymphoma non-specific, primary mediastinal B-cell lymphoma, grade 3b follicular lymphoma, indolent B-cell lymphoma (mantle cell lymphoma (MCL), marginal zone B-cell lymphoma (MZL)), slow lymphocytic transformed large B-cell lymphoma with previous treatment of anthracycline containing drugs and rituximab or other CD20 targeted therapies, that meets the criteria of the 2022 WHO classification of lymphoid tissue tumors. Adequate treatment with medication. Among them, inert B-NHL must have received at least 2 lines or more of standard treatment failure, while invasive B-NHL must have received at least 1 line or more of standard treatment failure. At least one regimen contains anti-CD20 monoclonal antibody monotherapy or combination therapy; Note: Relapse is defined as disease progression after sufficient treatment to achieve remission (CR or PR), with at least one regimen containing anti-CD20; Difficult to treat is defined as disease progression (PD or SD) within 6 months after full treatment with an anti-CD20 regimen without remission, or during the treatment period/after the end of full treatment;
4. At least one measurable tumor lesion. Measurable lesions (2014 Lugano lymphoma efficacy evaluation criteria): longest diameter of lymph nodes>15mm, extranodal lesions>10mm; lesions that have received local treatment such as radiotherapy before, if disease progression has been proven, are considered measurable lesions;
5. The ECOG score for physical fitness status ranges from 0 to 2 points;
6. Female or male participants of childbearing age should agree to have no fertility plans and take effective contraceptive measures within 6 months from the signing of the ICF until the last dose of the study drug is used;
7. Expected survival period is at least 3 months.

Exclusion Criteria:

1. Patients with current or previous primary central nervous system lymphoma (PCNSL) or secondary central nervous system involvement. Patients with central nervous system symptoms must undergo lumbar puncture and magnetic resonance imaging (MRI) examination to exclude them;
2. Patients who have received allogeneic hematopoietic stem cell transplantation and other organ transplantation, or who have received autologous hematopoietic stem cell transplantation within 100 days before the first dose;
3. Receive attenuated live vaccine within 4 weeks before the first administration or plan to receive it during the study period;
4. Patients with a history of malignant tumors within the past 5 years, except for those who have been completely cured of basal cell carcinoma of the skin or squamous cell carcinoma of the skin, melanoma in situ, and cervical carcinoma in situ, and/or any malignant tumor patients who have been cured without disease or have had no disease for at least 5 consecutive years;
5. Patients with active autoimmune diseases or a history of possible recurrence (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or high-risk patients. But the following patients may be considered for inclusion if the researchers assess disease stability: autoimmune hypothyroidism that only requires hormone replacement therapy; Skin diseases that do not require systemic treatment (such as eczema, rash that accounts for less than 10% of the body surface);
6. Patients who have undergone major surgery within 28 days prior to the first administration or are expected to undergo major surgery during the study period;
7. Subjects who require systemic corticosteroid treatment (>10mg/day prednisone or equivalent) or other immunosuppressive drugs within 7 days prior to the first administration or during the study period, but excluding topical corticosteroids via nasal spray, inhalation, or other routes, or systemic corticosteroids at physiological doses;
8. Subjects with active deep vein thrombosis or pulmonary embolism within the first 6 months of screening;
9. Patients currently suffering from interstitial lung disease or non infectious pneumonia, with active tuberculosis infection;
10. Systemic diseases not stably controlled after treatment, such as diabetes, serious organic cardiovascular and cerebrovascular diseases;
11. The patient's heart meets any of the following conditions: left ventricular ejection fraction (LVEF) ≤ 55%; New York Heart Association (NYHA) (see Appendix 3) Grade II or above congestive heart failure or active heart disease; Serious arrhythmias that require treatment (excluding atrial fibrillation and paroxysmal supraventricular tachycardia that have been determined by the researchers to have no impact on the trial); QTc interval ≥ 450ms for males and ≥ 470ms for females (QTc formula in Appendix 4); Within 6 months prior to administration, there has been a myocardial infarction or bypass or stent surgery; Other heart diseases deemed unsuitable for inclusion by researchers;
12. Human immunodeficiency virus (HIV) infection, hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) are positive during screening period, and HBV-DNA is higher than the normal range of the laboratory in the center; Patients who are positive for HCV antibodies during the screening period and have HCV-RNA levels higher than the normal range of the laboratory in their center;
13. Evidence of uncontrollable and severe active infections during screening (such as sepsis, bacteremia, mycosis, viremia, etc.);
14. Known subjects who have experienced severe allergic reactions to macromolecular protein preparations/monoclonal antibodies, as well as any components of the investigational drug in the past (CTCAE v5.0 grade ≥ 3);
15. Participated in clinical trials of other intervention drugs or medical devices within 4 weeks prior to the first administration of this study, or is currently undergoing treatment in other clinical trials (excluding non intervention studies);
16. Patients with a clear history of neurological or mental disorders, such as epilepsy, dementia, and poor compliance;
17. Pregnant or lactating women;
18. History of stroke or intracranial hemorrhage within 6 months;
19. Active or documented gastrointestinal bleeding within 6 months (such as esophageal or gastric varices, ulcer bleeding);
20. Researchers believe that patients who are not suitable to participate in the trial due to other reasons, such as rapid disease progression during the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | From day1 to day 21
  To evaluate the safety, tolerability, and determine the RP2D of IBR900 cell injection
The incidence and severity of adverse events (AEs) | From day 1 to day 30 after the last dose
  To evaluate the safety of IBR900 cell injection

SECONDARY OUTCOMES:
Complete response rate (CR) | From day 1 up to 9weeks
  The rate of subjects who achieved complete remission (CR) among all subjects
partial response rate (PR) | From day 1 up to 9weeks
  The rate of subjects who achieved partial remission (CR) among all subjects
objective response rate (ORR, including CR+PR) | From day 1 up to 9weeks
  The rate of subjects achieving CR and partial remission(PR) among all subjects
Duration of remission (DOR) | From day 1 up to disease recurrence ， progression or death because of any cause (maximun duration: 2.5 years ).
  Time from the subject's first assessment of the onset of remission to the first assessment of disease recurrence or progression or death from any cause
Overall survival (OS) | From day 1 up to death of any cause or follow-up loss (maximum duration : 4 years).
  Time from the start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Shanghai Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai